CLINICAL TRIAL: NCT01552694
Title: A Double Blind, Randomized, Placebo Controlled Study to Determine the Physiological Effectiveness of Januvia for Reducing Inflammation and Increasing EPC Number in HIV Infected Men and Women With Insulin Resistance and Central Adiposity.
Brief Title: Effectiveness of Sitagliptin for HIV Insulin Resistance and Inflammation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Kevin Yarasheski, PhD, Professor of Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 41052; 41052 (Other Grant/Funding Number: Merck)
Record Dates: First submitted 2012-03-08; First posted 2012-03-13 (Estimated); Results first posted 2015-03-05 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-03

CONDITIONS: Inflammation; Macrophage Infiltration; Cardiovascular Disease
Keywords: cardiometabolic complications
MeSH Terms: conditions — Inflammation; Cardiovascular Diseases | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin (Experimental): 100 mg sitagliptin/day for 2 months
  Interventions: Drug: Sitagliptin
- Placebo (Placebo Comparator): Matching placebo daily for 2 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin — Oral, 100 mg/day for 2 months
  Other Names: Januvia
  Arms: Sitagliptin
Drug: Placebo — oral, matching placebo daily for 2 months
  Arms: Placebo

SUMMARY:
People living with human immunodeficiency virus infection (HIV) have 2-4fold greater risk for developing diabetes and heart disease than the general population. They need safe and effective treatments that reduce the risk for developing diabetes and heart disease, and improve their quality of life. This project will explore whether a new anti-diabetes medication (Januvia) with a novel mechanism of action reduces inflammation, and improves blood vessel function in HIV infected men and women with several risk factors for developing cardiovascular disease.

DETAILED DESCRIPTION:
People living with human immunodeficiency virus (HIV+) infection have a 2-fold greater prevalence and incidence of T2DM and cardiovascular disease (CVD) than the general population. The investigators lack safe and effective treatments for these HIV related cardiometabolic complications despite the fact that HIV infected adults represent an ideal clinical population in which to study interactions among chronic low-grade pro-inflammatory processes that are linked to the development of adipose accumulation, insulin resistance, ß-cell secretory failure, vascular endothelial dysfunction, atherosclerosis and CVD. Dipeptidyl peptidase-IV (DPP4)-inhibitors represent a new drug class that safely and effectively regulate glycemia in T2DM, but have not been adequately tested in HIV. Of note, pre-clinical studies suggest that DPP4-inhibitors have several pleiotropic actions that may specifically benefit people living with HIV infection. For example, DPP4 inhibition reduced adipose macrophage infiltration & inflammation and increased the number of bone-derived endothelial progenitor cells in the circulation. Our preliminary findings indicate that DPP4 inhibition is virologically and immunologically safe in non-diabetic HIV+ adults taking combination antiretroviral therapy (in preparation), but the potential pleiotropic benefits have not been examined in HIV. The investigators propose a randomized, double blind, placebo controlled physiological study to test 2 potential pleiotropic benefits of DPP4 inhibition (100 mg sitagliptin/d, 8 wk): reduce circulating and adipose-specific markers of inflammation; and increase endothelial progenitor cell numbers used for vascular repair in 36 HIV+ adults with insulin resistance, central adiposity and CVD risk factors. The investigators hypothesize that sitagliptin will reduce circulating cytokine levels, reduce adipose tissue macrophage number and inflammation, and increase the number of circulating endothelial progenitor cells in HIV infected men and women. These physiological studies will advance our understanding about the efficacy of DPP4 inhibition in this high-risk group, and may help prevent the inexorable transition from insulin resistance to T2DM and CVD in HIV infected men and women.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 yr old HIV infected men and women.
* Stable (at least the past 6 months) on combined antiretroviral therapy (cART).
* Stable immune (> 300 CD4+ T-cells/µL) and virologic (< 50 copies HIV RNA/mL) status.
* Insulin resistant/impaired glucose tolerance (fasting glucose 100-125mg/dL, or 2-hr glucose 140-200mg/dL or fasting HOMA-IR= 2.5-6.0).
* Waist circumference > 102 cm (men), > 88 cm (women).
* BMI > 20 kg/m2.
* Fasting hypertriglyceridemia > 150 mg/dL.
* Low HDL-cholesterol (< 40 mg/dL in men or < 50 mg/dL in women).
* Platelet count > 30,000/mm3.
* Absolute neutrophil count > 750/mm3.
* Transaminases < 2.5x the upper limit of normal.
* Long-term non-progressors (not taking anti-HIV medications) are not eligible.

Exclusion Criteria:

* Diabetes (T2DM, IDDM or diabetic ketoacidosis) or taking any glucose-lowering medication (e.g., insulin, TZDs, metformin, sulfonylurea).
* Any agent that might artifactually alter glycemic control (e.g., glucocorticoids, megace, rhGH, GH-secretagogue, testosterone derivatives, creatine monohydrate, chromium picolinate, AA/protein supplements, medium- or long-chain fatty acids) during 6 months prior to or during enrollment.
* History of serious CV disease. NYHA Functional Class III or IV (e.g., recent MI, unstable angina, edema, CHF, CAD, CABG, stroke, resting hypertension > 160/95 mmHg), irregular heart rhythm, resting ST-segment depression > 1mm). Treatment with medications for CV condition (e.g., α- or ß-blockers). Some BP-lowering medications (Ca++channel blocker, diuretic, or ACE inhibitor) are permitted.
* Moderate to severe renal insufficiency. Serum creatinine > 1.7 mg/dL (men) > 1.5 mg/dL (women).
* Plan or anticipate a change in anti-HIV medications during the study.
* Lipid-lowering medications are permitted (fibrate or statin or niacin), but must be stable on that agent for at least 6 months prior to enrollment. Lipid-lowering agents cannot be started during the treatment period.
* Chronic hepatitis B (HBV-surface antigen positive). Active hepatitis C (detectable Hep C RNA).
* Positive urine drug test for opiates, methamphetamine, heroin, cocaine. Active substance abuse that the MD-scientist believes may compromise safety, compliance, interfere with study drug or data interpretation.
* Hematocrit < 34% in men or < 25% in women with symptoms (fatigue, "tired-legs", shortness of breath). Hemoglobin < 10 gm/dL with symptoms.
* Pregnant or nursing mothers. Women must agree to use an acceptable form of birth control during the study. If using birth control pills-must be stable on this medication for at least 6 months prior to enrollment.
* Active malignancy or treatment with chemotherapeutic agents or radiation therapy or any cytokine or anti-cytokine therapy during 6 months prior to enrollment.
* History of pancreatitis
* > 10% unintentional weight loss during the 6 months prior to enrollment.
* Reduced cognitive function/unable to provide voluntary informed consent. Prisoners are excluded.
* Blinded investigational drugs for 3 months prior to enrollment that will not be unblinded before enrollment.
* Nausea, vomiting, diarrhea (> 4 loose stools/day) that are unresponsive to treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-10; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin E Yarasheski, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Result] Best C, Struthers H, Laciny E, Royal M, Reeds DN, Yarasheski KE. Sitagliptin Reduces Inflammation and Chronic Immune Cell Activation in HIV+ Adults With Impaired Glucose Tolerance. J Clin Endocrinol Metab. 2015 Jul;100(7):2621-9. doi: 10.1210/jc.2015-1531. Epub 2015 May 4. PMID 25938633
- See also: Center for Clinical Studies- Washington University — https://ccs.wustl.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 38 participants were initially enrolled. 1 was lost to follow-up; 1 started a personal exercise training program while enrolled in the study. Any data collected on these 2 participants were excluded from the analysis. Both were initially enrolled in the placebo group.
Pre-assignment Details: 36 participants completed the trial with complete data.
Period: Overall Study
Arm/Group | Sitagliptin | Placebo
Started | 18 | 20
Completed | 18 | 18
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Placebo | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (9) | 52 (6) | 51 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 13 | 13 | 26
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 2 | 11 | 13
  African American | 16 | 7 | 23
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36
Weight [Mean (Standard Deviation); unit: kg] | 97 (21) | 102 (29) | 100 (25)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 32.7 (8.2) | 33.1 (8.2) | 32.9 (8.2)
Waist circumference [Mean (Standard Deviation); unit: cm] | 106 (19) | 112 (23) | 109 (22)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 124 (15) | 127 (14) | 125 (14)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 74 (9) | 78 (10) | 76 (10)
HIV duration [Mean (Standard Deviation); unit: years] | 14.9 (5.8) | 14.2 (7.5) | 14.6 (6.2)
CD4+ T-cell count [Mean (Standard Deviation); unit: cells/µL] | 731 (220) | 606 (218) | 668 (219)
CD8+ T-cell count [Mean (Standard Deviation); unit: cells/µL] | 1017 (542) | 801 (294) | 909 (418)

OUTCOME MEASURES:

1. Primary Outcome: Inflammatory Biomarker 1: Plasma hsCRP Concentration
Description: Fasting serum and plasma samples obtained at baseline and week 8 are batched for ELISA analysis (end of sudy) of hsCRP, IL-6 and D-dimer concentrations.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 18 | 18
mg/L
  Baseline | 3.4 (3.2) | 5.4 (4.5)
  Week 8 | 2.9 (2.6) | 7.4 (5.8)
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p = 0.006, t-test, 2 sided — A priori threshold for statistical significance was p<0.05. Unadjusted p-value compares the change (week 8 - baseline) for plasma hsCRP between the 2 groups

2. Primary Outcome: Inflammatory Biomarker 2: Plasma IL-6 Concentration
Description: There are 3 levels of the primary outcome measure; hsCRP, IL-6, and D-dimer concentrations measured at baseline and week 8
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 18 | 18
pg/mL
  Baseline | 1.36 (0.74) | 2.61 (1.91)
  Week 8 | 1.30 (0.55) | 2.65 (1.83)
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p = 0.24, t-test, 2 sided — A priori threshold for statistical significance was p<0.05. Unadjusted analysis

3. Primary Outcome: Inflammatory Biomarker 3: Serum D-dimer Concentration
Description: There are 3 levels of the primary outcome measure, hsCRP, IL-6, and D-dimer
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: µg FEU/mL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 18 | 18
µg FEU/mL
  Baseline | 0.32 (0.20) | 0.28 (0.15)
  Week 8 | 0.33 (0.24) | 0.31 (0.20)
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p = 0.78, t-test, 2 sided — A priori threshold for statistical significance was p<0.05. Unadjusted analysis

4. Secondary Outcome: Fold Change in Adipose Inflammation Marker CCL2 (MCP-1) mRNA Expression
Description: Adipose tissue from obese, insulin resistant subjects is characterized by increased macrophage infiltration and overexpression of inflammatory cytokines/chemokines. In adipose samples, mRNA expression for the macrophage inflammation marker CCL2 (MCP-1) was quantified. Fold change between population averages from baseline to 2 months for adipose macrophage CCL2 (MCP-1) mRNA expression is the outcome measure.
Time Frame: Baseline to 2 months
Population: Adipose tissue samples were not available from all participants. This secondary outcome includes fewer participants analyzed than the primary outcome.
Measure: Number; unit: fold change
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 11 | 7
fold change | -2.5 | -0.4

5. Secondary Outcome: Percent Change in Blood Endothelial Progenitor Cells
Description: Monocytes (PBMC) are isolated from 20 mL blood. CD34+/VEGFR2+/KDR+ monocytes represent cell markers for endothelial progenitor cells (EPC). CD34+/VEGFR2+/KDR+ monocytes are counted (flow cytometry) and expressed as a percentage of PBMC number. Percent change between population averages from baseline to 2 months for the EPC/PBMC ratio is calculated and reported as the outcome measure.
Time Frame: Baseline to 2 months
Population: CD34+/VEGFR2+/KDR+ monocytes (EPC) are a very rare cell type (<1% of PBMC). Not all blood samples contain EPC cells, or there are too few to count reliably. This measure was obtained in a subset of the total participants.
Measure: Number; unit: Percent change
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 12 | 11
Percent change | 0.3 | -0.2

ADVERSE EVENTS:
Arm/Group | Sitagliptin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/20
Other Adverse Events (participants affected / at risk) | 8/18 | 8/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=18) | Placebo (N=20)
Fatique, Fever, Chills, Loss of appetite, Weight Loss (General disorders) | 8 (9) | 7 (7) — All Other non-Serious Adverse Events under each organ system category were collected as a single event irrespective of the symptom.
Sinus, respiratoy urinary tract infections (Infections and infestations) | 2 (2) | 3 (3) — All Other non-Serious Adverse Events under each organ system category were collected as a single event irrespective of the symptom.
Rash, pruritus, easy bruising (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) — All Other non-Serious Adverse Events under each organ system category were collected as a single event irrespective of the symptom.
Chest pain, shortness of breath, wheezing, cough (Cardiac disorders) | 3 (3) | 4 (4) — All Other non-Serious Adverse Events under each organ system category were collected as a single event irrespective of the symptom.
Abdominal pain, nausea, vomiting, constipation, diarrhea, hypoglycemia (Gastrointestinal disorders) | 3 (3) | 6 (6) — All Other non-Serious Adverse Events under each organ system category were collected as a single event irrespective of the symptom.
Chnages in urinary frequency, painful urination, blood in urine (Renal and urinary disorders) | 2 (2) | 3 (3) — All Other non-Serious Adverse Events under each organ system category were collected as a single event irrespective of the symptom.
muscle ache, arthritis, swelling, weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5) — All Other non-Serious Adverse Events under each organ system category were collected as a single event irrespective of the symptom.
headaches, dizziness ,numbness, depression, anxiety, confusion (Nervous system disorders) | 4 (8) | 5 (10) — All Other non-Serious Adverse Events under each organ system category were collected as a single event irrespective of the symptom.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No